CLINICAL TRIAL: NCT02191436
Title: Psychosocial Factors and Adherence to Treatment in Patients With Hemophilia. A Multicenter Study
Brief Title: Adherence to Treatment in Hemophilia
Acronym: ADHERENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANA TORRES-ORTUÑO (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, ANA TORRES-ORTUÑO, PhD, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Other Study IDs: ADHERENCE; ADHE (Other: UMU)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Haemophilia
Keywords: Haemophilia; Adherence; Family Functioning; Quality of Life; Anxiety; Illness Behavior; Coping Strategies
MeSH Terms: conditions — Hemophilia A; Anxiety Disorders; Illness Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with haemophilia: Hemophilia patients (children, youth and adults) and parents of children with hemophilia under 18

SUMMARY:
Psychosocial factors and adherence to treatment in patients with hemophilia. A multicenter study. Multicenter cross sectional study of patients with hemophilia and their families

DETAILED DESCRIPTION:
Research project whose main objective is to assess adherence and major psychosocial issues affecting patients with hemophilia and their families treated at the Hematology and hemotherapy Services Clinical Hospital Universitario Virgen de la Arrixaca of Murcia and the University Hospital Carlos Haya, Malaga.

The data obtained in this project will identify those psychosocial aspects affecting patients and their families about the disease, its evolution and treatment of it. They will use different psychosocial questionnaires based on scientific evidence and the reliability of these, as well as its specific design for hemophilia patients. The main characteristics of the study are:

* Descriptive study of adherence to treatment of pediatric patients, adolescents and adults with hemophilia.
* Descriptive study of family functioning, perceived stress, anxiety and quality of life in parents of children with hemophilia under 14 years and adolescents with hemophilia, depending on the administered medical treatment, clinical and musculoskeletal patient situation.
* Descriptive study of illness behavior or perception of illness, perceived stress, anxiety, quality of life and coping strategies of young adults with hemophilia, depending on the medical treatment administered, and skeletal muscle clinical situation of the patient.
* Validation of psychosocial assessment tools in patients with hemophilia and their families.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A or B
* Patients followed at the Hematology Department of the hospitals included in the study
* Patients without cognitive disorders

Exclusion Criteria:

* Patients with other congenital coaguopatías
* Patients with more than 2 years without going to review your hospital
* Patients from other provinces of Spain

Ages: 6 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia treated at the Hospital Clínico Universitario Virgen de la Arrixaca de Murcia, and the Hospital Clínico Universitario Carlos Haya (Málaga)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-11 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Assess the perception of quality of life | Screening visit
  The quality of life assessed with the questionnaires: Short Form-36 Health Survey (SF-36) and A36 Hemofilia-QoL for adults; and Child Report Form (CHIP-CE) and Haemo-QoL, for children.
Assess the perception of illness of the patients | Screening visit
  To measure this variable we use the Illness Perception Questionnaire Revised (IPQ-R).
Assess anxiety of patients and parents of children with hemophilia. | Screening visit
  To evaluate this variable we use the State-Trait Anxiety Inventory (STAI)
To assess illness behavior of patients. | Screening visit
  To assess this variable we use the illness behaviour questionnaire (IBQ).
Assessing coping strategies of patients. | Screening visit
  To assess this variable we use the Coping Scale questionnaire.
Assess the perception of family functioning of parents of children with hemophilia | Screening visit
  To assess this variable we use the Family Functioning Evaluation Scale (FACES III).
Assess the perceived stress of parents of children with hemophilia. | Screening visit
  To assess this variable we use the Pediatric Inventory for Parents (PIP).
Assessing the personality traits of children with hemophilia. | Screening visit
  To assess this variable we use the Eysenck Personality Questionnaire Junior (EPQ-J)
Assess adherence to treatment of patients with hemophilia. | Screening visit
  To assess this variable we use the Beliefs About Medication Questionnaire (BMQ).

SECONDARY OUTCOMES:
Assess the clinical data of the patient | Screening visit
  Type of hemophilia (A or B), severity of hemophilia (severe, moderate or mild), treatment type (a demand or prophylaxis), presence of ingibidores, history of hemarthrosis, dosage factor VIII / IX
Assess the demographic data of the patient | Screening visit
  Age, history of hemophilia in the family, marital status (single, married, divorced), education (university, basic), employment status (unemployed, self-employed, employed by others), distance to hospital

CONTACTS AND LOCATIONS:
Overall Officials: RUBÉN CUESTA-BARRIUSO, PhD, Principal Investigator — UNIVERSIDAD CATÓLICA SAN ANTONIO, MURCIA
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia, Spain